CLINICAL TRIAL: NCT07390643
Title: Determining ImpactS of Multi-Cancer Early detectiOn Tests oVER Time in Symptomatic Patients: The DISCOVER Study
Brief Title: The DISCOVER Study
Acronym: DISCOVERY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Elizabeth ODonnell, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 25-467
Record Dates: First submitted 2026-01-26; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Cancer Diagnosis
Keywords: Cancer; Cancer Diagnosis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Galleri MCED Test (Experimental): Enrolled participants will complete:
  * Baseline visit with blood draw and questionnaires
  * Return of test results:
    * For a positive result, diagnostic work-up could include clinic visits, biopsy, surgery, imaging assessments such as ultrasound, Computed Tomography (CT) scans, or Magnetic Resonance Imaging (MRI) scans. If standard, diagnostic work-up is positive or negative for cancer, follow up will be at the discretion of the principal investigator.
    * For a negative MCED blood test with standard, diagnostic work-up that is negative, follow-up will be at the discretion of the principal investigator.
  * Online post-test questionnaire
  * Online post-diagnostic questionnaire
  * Follow up will be up to 24 months
  Interventions: Device: GRAIL Galleri MCED test

INTERVENTIONS:
Device: GRAIL Galleri MCED test — A multi-cancer early detection (MCED) blood test.

SUMMARY:
The purpose of this research study is to evaluate the possible benefits of screening with an investigational, but commercially available blood test designed to detect many types of cancer.

The name of the screening blood test being studied is:

-GRAIL Galleri MCED test

DETAILED DESCRIPTION:
The purpose of this pilot research study is to evaluate the possible benefits of screening with an investigational, but commercially available blood test designed to detect many types of cancer. "Investigational" means that this test is being studied and is not approved or cleared by the Food and Drug Administration (FDA).

The multi-cancer early detection test looks for small pieces of genetic material, called DNA (deoxyribonucleic acid), in the blood that may indicate the presence of cancer, and the test may also be able to suggest what type of cancer is present.

The research study procedures include screening for eligibility, in-clinic visit, blood tests, and questionnaires.

It is expected that about 110 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 22 years old
* Have signs and symptoms suggestive of cancer and/or have imaging related to signs and symptoms of cancer being evaluated in the Cancer Diagnostic Service clinic

Exclusion Criteria:

* Individuals diagnosed with invasive malignancy within 3 years of enrollment
* Individuals with active cancer requiring active therapeutic intervention at the time of participation (hormone therapy for breast/prostate cancer is considered acceptable and will not preclude participation)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Multi-cancer Early Detection (MCED) Positive Cancer Type | MCED testing will be performed at enrollment, with diagnostic resolution and cancer type determination expected within 12 months.
  MCED positive cancer type is defined as the type of cancer detected by the MCED test. Cancer type will be defined and recorded using ICD-O-3 codes for primary anatomic site (topography) and histology (morphology).
Multi-cancer Early Detection (MCED) Positive Cancer Incidence | MCED testing will be performed at enrollment, with diagnostic resolution and cancer type determination expected within 12 months.
  MCED positive cancer incidence is defined as the number of cancers detected by the MCED test.
Multi-cancer Early Detection (MCED) Positive Cancer Stage | MCED testing will be performed at enrollment, with diagnostic resolution and cancer type determination expected within 12 months.
  MCED positive cancer stage is defined as the stage of cancer detected by the MCED test.
Multi-cancer Early Detection (MCED) Undetected Cancer Type | MCED testing will be performed at enrollment, with diagnostic resolution and cancer type determination expected within 12 months.
  MCED undetected cancer type is defined as the cancer type detected by standard diagnostic methods that was not identified by the MCED test. Cancer type will be recorded using ICD-O-3 codes for both the primary anatomic site (topography) and histology (morphology).
Multi-cancer Early Detection (MCED) Undetected Cancer Incidence | MCED testing will be performed at enrollment, with diagnostic resolution and cancer type determination expected within 12 months.
  MCED undetected cancer incidence is defined as the number of cancers detected by standard diagnostic methods that was not identified by the MCED test.
Multi-cancer Early Detection (MCED) Undetected Cancer Stage | MCED testing will be performed at enrollment, with diagnostic resolution and cancer type determination expected within 12 months.
  MCED undetected cancer stage is defined as the stage of cancer detected by standard diagnostic methods that was not identified by the MCED test. Hodgkin lymphoma (HL) is typically staged using the Ann Arbor system; non-Hodgkin lymphoma (NHL) is staged according to the Lugano classification; multiple myeloma (MM) is staged using the International Staging System (ISS); and chronic lymphocytic leukemia (CLL) is staged according to the Rai staging system.

SECONDARY OUTCOMES:
Positive Predictive Value (PPV) of Multi-cancer Early Detection (MCED) | 12 months
  PPV of the MCED test will be calculated as the proportion of participants diagnosed with cancer among all participants who had positive MCED test results.
Number of Additional Tests | MCED testing will be performed at enrollment, with diagnostic resolution and cancer type determination expected within 12 months.
  Number of additional tests is defined as total number of diagnostic tests performed to achieve final diagnostic resolution after the initial MCED test.
Types of Additional Tests | MCED testing will be performed at enrollment, with diagnostic resolution and cancer type determination expected within 12 months.
  Types of additional tests are defined as the specific types of diagnostic tests performed to reach final diagnostic resolution after the initial MCED test.
Tissue of Origin Correct Prediction Rate | MCED testing will be performed at enrollment, with diagnostic resolution and cancer type determination expected within 12 months.
  Tissue of origin correct prediction rate is defined as the proportion of participants in whom the tissue of origin predicted by the GRAIL Galleri® MCED test matches the confirmed cancer site, based on cancer status assessments.
Qualitative Provider Assessment of MCED Test Utility | 24 months
  At the end of the study, participating providers will be surveyed to assess their attitudes, perceptions, and experiences regarding the utility and integration of MCED tests in clinical practice. The assessment includes multiple-choice questions, and open-ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth O'Donnell, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu